CLINICAL TRIAL: NCT05680506
Title: Effects of Pain Neuroscience Education With Conventional Physical Therapy in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/21
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of two groups. One will recieve conventional physcial therapy only and the second will recieve conventional physcial therapy with pain neuroscience education.Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the particpant belong to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education group (Experimental): Pain neuroscience education 10- 15min Hot pack(10 min) TENS Kaltenborn Moilization technique at L4-L5 segment stretchings and stabilization exercises. (5 reps/1 set) Total duration:40 min/session
  Interventions: Procedure: Pain neuroscience education; Procedure: Standard Therapy
- Standard therapy group (Active Comparator): Hot pack(10 min) TENS Kaltenborn Mobilization technique at L4-L5 segment stretchings and stabilization exercises (5 reps /1 set) Total duration:30 min/session
  Interventions: Procedure: Standard Therapy

INTERVENTIONS:
Procedure: Pain neuroscience education — Pain neuroscience education will be given in form videos,pictures, stories and metaphors for 2 times per week for 4 weeks.
  Arms: Pain neuroscience education group
Procedure: Standard Therapy — Hot pack,TENS, Kaltenborn grade 1 and 2 mobilizations, stretchings and lumbar stabilization exercises

SUMMARY:
Low back pain is currently considered to be the most common cause of disability.When low back pain occurs sensitivity of body increases which decreases overall body activity.Physical inactivity negatively effects recovery from chronic low back pain.Patients with chronic low back pain experience psychological anxiety and depression which leads to fear of pain and movement.There are various treatment options for chronic low back pain.But most treatment options deal with biomedical aspect of disease.Pain neuroscience education deals with psychological aspect of disease.By combining both treatment options we will be able to evaluate the combined biopsychosocial aspect of treatment.This study will mainly focus on the education of patients regarding neuroscience be hind their chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is currently considered to be the most common cause of disability.This is the single greatest cause of years lived with disability.When low back pain occurs the sensitivity of body increases which decreases overall body activity.Physical inactivity negatively effects recovery from chronic low back pain.Patients with chronic low back pain experience psychological anxiety and depression which leads to fear of pain and movement. There are various treatmet options for chronic low back pain.But most treatment options deal with biomedical aspect of disease.Pain neuroscience education deals with psychological aspect of disease.By combining both treatment options we will be able to evaluate the combined biopsychosocial aspect of treatment.This study will mainly focus on education of patients regarding neuroscience behind their chronic low back pain.

A randomized control trial will be conducted in Tariq Memorial Neuro Clinic Islambad using non-probability purposive sampling.Participants will be briefed regarding the study objectives, procedure, risks and benefits of treament, voluntary participation and right to withdraw.Written informed consent will be taken from all the participants before conducting the research.Details of exercise program will be explained to them.Patients wiith chronic low back pain will be reffered by neuro-physician.Screening will be done by using Keel Start Back screening tool.Then the selected participants will be randomized into 2 groups(experimental group and control group)via sealed envelope method. Participants will complete Numeric Rating Pain Scale(NRPS) for pain, Roland Morris Disability Questionnaire for disability measurement and Tampa Scale for kinesiophobia.All of these measurements will be taken at baseline and then after 4 weeks of intervention.

The treatment protocol of both groups is as follows:

Group 1(Control group):hot pack, TENS for 15 mins, mobilization at L4-L5 segment, stretchings and stabilization exercises (5 reps/1set) Group 2(Experimental group):Pain neuroscience education for 15 mins, hot pack, TENS,mobilization at L4-L5 segment, stretchings and stabilization exercises.(5 reps/1 set)

ELIGIBILITY:
Inclusion Criteria:

* Both male and female of age 40-65 years
* Patients with chronic primary low back pain (medium risk patients on Start Back Screening Tool)

Exclusion Criteria:

* patients with motor and sensory dysfunction
* patients with neurological abnormalities and muscle paalysis
* patients with dizziness and uncontrolled hypertension
* patients who could not take the basic posture of lumbar stabilization exercises because of pain

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured on numeric rating pain scale. It consists of 11 points( interval 0-10), where 0 corresponds to no pain and 10 corresponds to worst pain imaginable. A graphical representation of 11 spaces is used for patients own evaluation of his or her pain
Disability | 4 weeks
  The activity disorder index is assessed using the Roland Morris Disability Questionnaire RMDQ. It consists of 0-24 point scale. The score ranges from 0 (no disability) to 24 (maximum disability).
Kinesiophobia | 4 weeks
  Tampa scale is used in patients with chronic musculoskeletal pain.It composed of 17 items scoring range from 1-4: (1) strongly disagree, (2) disagree, (3) agree,(4) strongly agree. For items 4,8,12 and 6 its vice versa.The total score of scale range from 17-68, where 17 means no kinesiophobia, 68 means severe kinesiophobia and 37 means there is kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan